CLINICAL TRIAL: NCT05232708
Title: A Study to Demonstrate Bioequivalence Between Semaglutide Formulation for the DV3396 Pen-injector and the Formulation for the PDS290 Semaglutide Pen-injector
Brief Title: A Clinical Trial Looking at the Comparability of 2 Different Forms of Semaglutide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-4885; 2021-003216-25 (EudraCT Number); U1111-1266-4076 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-01-17; First posted 2022-02-10 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteers (Diabetes Mellitus, Type 2)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide B, 1.34 mg/mL followed by Semaglutide D, 1.0 mg/mL (Experimental)
  Interventions: Drug: Semaglutide B, 1.34 mg/mL; Drug: Semaglutide D, 1.0 mg/mL
- Semaglutide D, 1.0 mg/mL followed by Semaglutide B, 1.34 mg/mL (Experimental)
  Interventions: Drug: Semaglutide D, 1.0 mg/mL; Drug: Semaglutide B, 1.34 mg/mL

INTERVENTIONS:
Drug: Semaglutide B, 1.34 mg/mL — Subjects will receive single dose of 0.5 mg Semaglutide B, 1.34 mg/mL subcutaneously.
  Arms: Semaglutide B, 1.34 mg/mL followed by Semaglutide D, 1.0 mg/mL
Drug: Semaglutide D, 1.0 mg/mL — Subjects will receive single dose of 0.5 mg Semaglutide D, 1.0 mg/mL subcutaneously.
  Arms: Semaglutide B, 1.34 mg/mL followed by Semaglutide D, 1.0 mg/mL
Drug: Semaglutide D, 1.0 mg/mL — Subjects will receive single dose of 0.5 mg Semaglutide D, 1.0 mg/mL subcutaneously.
  Arms: Semaglutide D, 1.0 mg/mL followed by Semaglutide B, 1.34 mg/mL
Drug: Semaglutide B, 1.34 mg/mL — Subjects will receive single dose of 0.5 mg Semaglutide B, 1.34 mg/mL subcutaneously.
  Arms: Semaglutide D, 1.0 mg/mL followed by Semaglutide B, 1.34 mg/mL

SUMMARY:
In this trial, two approved solutions of the medicine semaglutide will be compared in healthy volunteers. The purpose of this trial is to see if semaglutide B and semaglutide D solutions are comparable with regards to moving into, through and out of the body when given in two separate injections. Participants will receive semaglutide B and semaglutide D in different periods of the trial (Period 1 and Period 2). Participants will receive 1 subcutaneous injection of semaglutide B (0.5 mg) and 1 subcutaneous injection of semaglutide D (0.5 mg). The trial will last for 87 to 120 days (about 3 to 4 months), depending on how long the screening period (2 to 28 days) and washout period (14 to 21 days) are. Participants will have a screening visit, followed by an in house stay (5 nights/6 days) and 9 visits for each period. Participants will have to fast for at least 6 hours overnight with only water allowed before receiving the trial medicine on the second day of in house stay (Day 1) in Period 1 and Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 20-55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 25.0 and 34.9 kilogram per meter square (kg/m^2) (both inclusive)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive method
* Any disorder which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol
* Use of prescription medicinal products or non-prescription drugs, except routine vitamins, topical medications, highly effective contraceptives and occasional use of paracetamol and acetylsalicylic acid, within 14 days prior to the day of screening
* Abuse or intake of alcohol, defined as any of the below:

  * Known or suspected alcohol abuse within 1 year before screening (defined as regular intake of more than an average intake of 24 grams (g) alcohol daily for men and 12 g alcohol daily for women - 12 g of alcohol equals about 300 milliliters (mL) of beer or lager, 100 mL of wine, or 25 mL spirits).
  * Positive alcohol test at screening.
* Abuse or intake of drugs, defined as any of the below:

  * Known or suspected drug or chemical substance abuse within 1 year before screening
  * Positive drug of abuse test at screening

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
AUC0-last,sema 0.5mg: Area under the semaglutide concentration-time curve from time 0 until last quantifiable measurement after single dose of s.c. semaglutide 0.5 mg | 0-840 hours after a single dose of s.c. semaglutide 0.5 mg
  Measured in h*nmol/L
Cmax,sema,0.5mg: maximum observed semaglutide concentration-time after single dose of s.c. semaglutide 0.5 mg administration | 0-840 hours after a single dose of s.c. semaglutide 0.5 mg
  Measured in nmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Parexel CPRU, Level 7, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com